CLINICAL TRIAL: NCT05900791
Title: Incidence of Persistent Pain After Knee Arthroplasty: A Nationwide Cross-sectional Survey Study
Brief Title: Persistent Pain After Knee Replacement
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Jens Laigaard, Principal investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: P-2023-4
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Persistent Postsurgical Pain; Arthritis Knee; Neuropathic Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Primary knee arthroplasty — All patients surveyed have undergone primary knee arthroplasty approximately 1 year prior to survey distribution
  Other Names: Primary knee replacement

SUMMARY:
This study is a nationwide cross-sectional survey on pain and satisfaction after knee arthroplasty (KA). Please find the full protocol uploaded at ClinicalTrials.gov

The goal of this observational study is to study pain and satisfaction in patients operated with knee arthroplasty. The main question it aims to answer are:

* What is the incidence of persistent postsurgical pain in unselected knee arthroplasty patients
* What is the level of satisfaction in unselected knee arthroplasty patients?

Participants will be asked to answer a 22-item questionnaire.

DETAILED DESCRIPTION:
The study is registered at the Capitol region of Denmark's regional research listing (Pactius) with identifier P-2023-4, approved 4 January 2023. The resulting paper will be reported according to the CROSS checklist for standardised reporting of survey studies. Wherever needed, a trained linguist translated questions from English to Danish and vice versa. The Danish and an English version of the questionnaire will be available in the final publication.

* Study design: This study is a nationwide cross-sectional survey.
* Patient involvement: A panel of KA patients helped develop the questionnaire, i.e., testing and selecting the questions.
* Questionnaire: The questionnaire is composed of 22 questions (please see the uploaded protocol), however patients answering "No" to question 3 skips questions 4-17 concerning pain in the operated knee. Only question 3, 4, 20, and 21 are mandatory as to avoid non-respondents. The full questionnaire translated to English can be found in the supplementary material in the protocol. Contact information for the first author (JL) is supplied in the contact letter in case the patients have difficulties with filling in the questionnaire, have questions, or believe they have been selected mistakenly. Similar or identical questions to those in a survey published in 2006 to increase the ability to compare results (i.e., questions 3-5, 8, 10 and 18)
* Sample characteristics: Eligible patients are all adult (18 years or older) patients operated with primary total or medial unicompartmental KA for osteoarthritis between August 1 and November 30, 2023. Legally incompetent citizens, i.e., persons with a legal guardian, will not be asked to participate. For total KA, patients are identified from the Danish National Patient Register through the Danish Health Data Authority (SKS-code DM17 [knee osteoarthritis] + KNGB20, KNGB30 or KNGB40 [primary total knee arthroplasty]). For medial unicompartmental KA, patients are identified from the Danish National Patient Register through the Danish Health Data Authority (SKS-code DM17 [knee osteoarthritis] + KNGB01 or KNGB11 [primary medial unicompartmental knee arthroplasty]).
* Sample size calculation: The sample size calculation is based on the primary outcome in total KA patients. With an estimated 16% incidence of the primary outcome3 and a 70% response rate, 3172 patients are needed to yield a 95% confidence interval of 3 percentage points (14.6-17.6). In our opinion, this level of certainty is appropriate because differences less than this, may be hard to interpret by clinicians and patients. Sampling patients that were operated during 4 months outside holiday season should yield approximately this number of identified patients
* Ethical considerations: The local institutional review board approved the study, and the Danish Health Data Authority will provide contact information for potential respondents. Telephone numbers for non-respondents are found by searching the CPR number in the electronic patient files, but without accessing the patients' health data. According to Danish legislation, approval from the national ethics committee is neither required nor possible to obtain for survey studies.

ELIGIBILITY:
Inclusion Criteria:

- Patients operated with primary knee arthroplasty for osteoarthritis 12-15 months before survey distribution

Exclusion Criteria:

- Legally incompetent citizens, i.e., persons with a legal guardian, will not be asked to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For total KA, patients are identified from the Danish National Patient Register through the Danish Health Data Authority (SKS-code DM17 [knee osteoarthritis] + KNGB20, KNGB30 or KNGB40 [primary total knee arthroplasty]).
  For medial unicompartmental KA, patients are identified from the Danish National Patient Register through the Danish Health Data Authority (SKS-code DM17 [knee osteoarthritis] + KNGB01 or KNGB11 [primary medial unicompartmental knee arthroplasty]).
Sampling Method: Non-Probability Sample
Enrollment: 3710 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Moderate/Severe persistent postsurgical pain | 11-15 months postsurgically
  The main outcome is the number of patients with moderate or severe persistent postsurgical pain in the operated knee, defined as patients with a numerical rating scale (NRS) score higher than 3. The NRS score was dichotomised for the primary outcome because this is more intuitively understood by patients and clinicians. This outcome will be reported as percentage of all patients with 95% confidence interval, which is calculated with assumed binomial distribution as p ± 1.96 √( (p (1 - p) ) / n)

SECONDARY OUTCOMES:
How satisfied are you with the outcome of your knee replacement surgery? Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied, Very dissatisfied | 11-15 months postsurgically
  Reported as n (%) for each response option. The 1st question assesses overall satisfaction with surgery and have been translated directly from the questionnaire used by the Swedish Arthroplasty Register.
Knowing what your knee replacement surgery did for you, if you could go back in time, would you still have undergone this surgery? Yes, No, Uncertain | 11-15 months postsurgically
  Reported as n (%) for each response option.
Pain frequency: Do you still have pain in the operated knee? Yes, constantly; Yes, daily; Yes, a few times a week; Yes, more rarely; No | 11-15 months postsurgically
  Reported as n (%) for each response option.
Numerical Rating Scale (NRS) pain: Please rate your pain in the operated knee by indicating the number that best describes your pain on average during the last week. 0 means 'No pain' and '10' means 'Pain as bad as you can imagine'. | 11-15 months postsurgically
  Reported as median (interquartile range [IQR]) and number of respondents
Pain domain of the likert-scale version 3.1 of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). | 11-15 months postsurgically
  The five questions in the WOMAC pain domain can be scored 0-4, where 0 is 'none' and 4 is 'extreme'. This results in an overall score of 0-20, which will be reported as median (IQR). Moreover, each response option of the individual questions are reported as n (%).
Pain interference: In total, how much does the pain in the operated knee bother you in your everyday life? Not at all, A little, Some, Much, Very Much | 11-15 months postsurgically
  Reported as n (%) for each response option
Douleur Neuropathique 4 questions (DN4) interview | 11-15 months postsurgically
  Each of the seven questions in the DN4 interview can be scored 0/1 (no/yes), which results in an overall score of 0-7. A score ≥3 constitutes 'possible' neuropathic pain. Both the median (IQR) DN4 interview score and number of patients (% of all patients) with possible neuropathic pain will be reported.
Other pain: Do you have chronic pain, other than from your operated knee? Yes; No. [If yes] -> Please describe your pain condition | 11-15 months postsurgically
  Pain conditions will be categorised independently by two authors and reported as n (%).
Analgesic use: Do you take analgesic medication(s) daily or almost daily? Yes; due to pain in the operated knee; Yes, due to other pain; No. [If yes] -> Which medication(s)?: | 11-15 months postsurgically
  Reported as n (%).
Height (cm) | 11-15 months postsurgically
Weight (kg) | 11-15 months postsurgically

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, MD, PhD, Professor, Study Director — Department of orthopedic surgery, Bispebjerg University Hospital, Denmark
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The full dataset will be stored at the Danish national archive (www.rigsarkivet.dk) if possible

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05900791/Prot_SAP_000.pdf